CLINICAL TRIAL: NCT02087150
Title: A Randomized Clinical Study of Safety and Efficacy for the Eustachian Tube Balloon Catheter (ELLIOTT)
Brief Title: Study of Safety and Efficacy for the Eustachian Tube Balloon Catheter
Acronym: ELLIOTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPR005029
Record Dates: First submitted 2014-03-06; First posted 2014-03-14 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Eustachian Tube Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Medical management (MM) (No Intervention): Medical management will consist of 6 weeks of daily intranasal steroid (triamcinolone acetonide)
- Eustachian tube balloon catheter (ETBC) plus MM (Experimental): Eustachian tube dilation with the ETBC plus medical management
  Interventions: Device: Acclarent Eustachian Tube Balloon Catheter (ETBC)

INTERVENTIONS:
Device: Acclarent Eustachian Tube Balloon Catheter (ETBC)
  Arms: Eustachian tube balloon catheter (ETBC) plus MM

SUMMARY:
The objective of this study is to determine whether Eustachian tube dilation in conjunction with medical management or medical management alone is effective for treating Eustachian tube dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female aged 22 years and older
* Persistent Eustachian tube dysfunction
* Failure of medical management
* Positive diagnosis of ETD
* Absence of internal carotid artery (ICA) dehiscence
* Able to read and understand English

Exclusion Criteria:

* Females who are pregnant or lactating
* Anatomy that requires an adjunctive surgical procedure
* Concomitant nasal or sinus procedures planned on the same day as surgical procedure
* Concomitant ear procedures planned on the same day as surgical procedure
* History of major surgery of the head or neck within four (4) months prior to surgery
* History of patulous ET
* History of fluctuating sensorineural hearing loss
* Active acute otitis media
* Tympanic membrane perforation
* Tympanosclerosis
* Acute upper respiratory infection
* Temporomandibular joint disorder
* Cleft palate
* Craniofacial syndrome
* Cystic fibrosis
* Ciliary dysmotility syndrome
* Systemic mucosal or immunodeficiency disease
* Intolerance of medication for ETD
* Prior intervention of Eustachian tube

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Poe, MD, PhD, Principal Investigator — Boston Children's Hospital; Vijay Anand, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center and Weill Medical College of Cornell University
Locations (21):
- United States (21):
  - California Ear Institute, East Palo Alto, California
  - George Washington Medical Faculty Associates, ENT Center, Washington D.C., District of Columbia
  - ENT of South Florida, Boca Raton, Florida
  - ENT of South Florida, Boynton Beach, Florida
  - Florida Ear & Sinus Center, Sarasota, Florida
  - ENT of Georgia, Atlanta, Georgia
  - Piedmont Ear, Nose & Throat &Related Allergy, Atlanta, Georgia
  - Witham Health Services, Lebanon, Indiana
  - Red River Sinus Center, Alexandria, Louisiana
  - Our Lady of the Lake Hospital, Baton Rouge, Louisiana
  - Children's Hospital, Boston, Massachusetts
  - Health Partners Specialty Center, Saint Paul, Minnesota
  - The Sinus Center of the South, Ocean Springs, Mississippi
  - Vijay Anand, LLC, New York, New York
  - Ear, Nose, Throat and Allergy Associates, LLP, Port Jefferson, New York
  - Ear, Nose, Throat and Allergy Associates, LLP, White Plains, New York
  - Charlotte Eye, Ear, Nose &Throat Associates, Charlotte, North Carolina
  - Carolina Ear and Hearing Clinic, Raleigh, North Carolina
  - Texas Healthcare, PLLC, Fort Worth, Texas
  - Ear Medical Group, San Antonio, Texas
  - Meriter Monona, Monona, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
A publication is planned

REFERENCES:
- [Derived] Swords C, Smith ME, Patel A, Norman G, Llewellyn A, Tysome JR. Balloon dilatation of the Eustachian tube for obstructive Eustachian tube dysfunction in adults. Cochrane Database Syst Rev. 2025 Feb 26;2(2):CD013429. doi: 10.1002/14651858.CD013429.pub2. PMID 40008607

RESULTS

PARTICIPANT FLOW:
Groups:
- Lead-In: Subjects enrolled in Lead-In Group
- Randomized ETBC: Subjects enrolled and randomized to treatment with the Eustachian Tube Balloon Catheter (ETBC) plus Medical Management (MM)
- Randomized MM: Subjects enrolled and randomized to treatment with medical management (MM) only. Subjects randomized to the MM arm were allowed the option to cross-over to have a procedure with the ETBC after completion of the 6 week follow-up visit. Cross-over subject were followed to 12 weeks post-procedure only. Thereafter, they were exited from the study and not required to undergo the 24 week and 52 week follow-up visits
Period: Overall Study
Arm/Group | Lead-In | Randomized ETBC | Randomized MM
Started | 81 | 162 | 80
Had a Lead-in or Randomized ETBC Proc | 80 | 149 | 0
Received a Crossover MM ETBC Procedure | 0 | 0 | 70
Completed | 71 | 128 | 69
Not Completed | 10 | 34 | 11
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 6 | 13 | 7
Not completed — Withdrawal by Subject | 2 | 5 | 3
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Procedure not done | 1 | 13 | 0
Not completed — F/U not completed w/in study window | 0 | 0 | 1
Not completed — Other | 1 | 0 | 0
Not completed — Pt moved out of town | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lead-In | Randomized ETBC | Randomized MM | Total
Number analyzed (Participants) | 81 | 162 | 80 | 323
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.7 (14.1) | 55.6 (14.3) | 57.7 (13.4) | 55.6 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 77 | 48 | 155
  Male | 51 | 85 | 32 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 9 | 2 | 12
  Not Hispanic or Latino | 80 | 153 | 78 | 311
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 12 | 8 | 23
  White | 77 | 147 | 67 | 291
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Analysis: Number of Randomized Subjects With Tympanogram Normalization at 6 Weeks
Description: The primary efficacy analysis compares randomized subjects with tympanogram normalization (Types B or C normalized to Type A) in all indicated ears at 6 weeks in the investigational arm versus the control arm. Per protocol, tympanogram types are defined as follows: Type A: Peak compliance occurs between +50 and -100 daPa, with minimum peak height of 0.2ml. Indicates NORMAL middle ear function Type B: No sharp peak and a rounded line. Indicates ABNORMAL middle ear function Type C: Peak compliance occurs beyond -100 daPa. Indicates ABNORMAL middle ear function
Time Frame: 6 Week Follow-Up Visit
Population: Primary Analysis Cohort (PAC): The PAC is defined as all randomized subjects who receive a study treatment for which they are randomized and have completed their primary analysis visits (i.e. completer analysis with baseline and 6 week tympanogram).
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized ETBC | Randomized MM
Number analyzed (Participants) | 143 | 72
Participants | 73 | 10

2. Secondary Outcome: Secondary Efficacy Endpoint: Number of Randomized Subjects With MID Improvement From Baseline of 0.5 Points or More at 6 Weeks
Description: The secondary efficacy endpoint will consist of comparison of subjects achieving at least a minimally important difference (MID) level improvement of 0.5 points on the ETDQ-7 at 6 weeks post-treatment in the investigational arm versus the proportion of subjects achieving at least an MID level improvement on the ETDQ-7 at 6 weeks post-randomization in the control arm The ETDQ-7 is a seven-item ETD specific validated quality of life survey. A mean item score of greater or equal to 2.1 indicates the presence of ETD.
Time Frame: 6 Week Follow-Up Visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized ETBC | Randomized MM
Number analyzed (Participants) | 143 | 72
Participants | 128 | 32

3. Other Pre Specified Outcome: Exploratory Endpoint: Number of Randomized Subjects With Normalized Tympanometry at 12.24,52 Weeks
Description: Evaluation of subjects experiencing normalization of tympanometry at 12 weeks, 24 weeks, and 52 weeks post-treatment in the investigational arm and evaluation of subjects experiencing normalization of tympanometry at 12 weeks, 24 weeks, and 52 weeks post-randomization in the control arm. As MM subjects were allowed to receive a crossover procedure after their 6-week follow-up visit, there is a limited number of MM subjects who completed the 12/24/52 visits.
Time Frame: 12, 24, 52 Week Follow-Up
Population: Per-Protocol Cohort: All randomized subjects expect those who: • Did not complete a baseline or respective follow-up assessment for the time point under analysis • Did not receive the treatment for which they were randomized • Had any major protocol deviation(s)
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized ETBC | Randomized MM
Number analyzed (Participants) | 149 | 80
Participants
  12 Week Visit: number analyzed (Participants) | 136 | 17
  12 Week Visit | 64 | 7
  24 Week Visit: number analyzed (Participants) | 134 | 9
  24 Week Visit | 78 | 5
  52 Week Visit: number analyzed (Participants) | 128 | 4
  52 Week Visit | 71 | 2

4. Other Pre Specified Outcome: Exploratory Endpoint: Number of Randomized Subjects With ETDQ-7 Improvement at 12, 24, 52 Weeks
Description: Evaluation of subjects achieving at least a MID level improvement of 0.5 points at 12 weeks, 24 weeks, and 52 weeks post-treatment in the investigational arm and evaluation of subjects achieving at least a MID level improvement at 12 weeks, 24 weeks, and 52 weeks post-randomization in the control arm. As MM subjects were allowed to receive a crossover procedure after their 6-week follow-up visit, there is a limited number of MM subjects who completed the 12/24/52 visits.
Time Frame: 12,24,52 Week Follow-Up Visit
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized ETBC | Randomized MM
Number analyzed (Participants) | 149 | 80
Participants
  12 Week Visit: number analyzed (Participants) | 134 | 15
  12 Week Visit | 118 | 9
  24 Week Visit: number analyzed (Participants) | 134 | 9
  24 Week Visit | 123 | 5
  52 Week Visit: number analyzed (Participants) | 124 | 4
  52 Week Visit | 111 | 3

5. Other Pre Specified Outcome: Exploratory Endpoint: WPAI at 6,12,24,52 Weeks
Description: Evaluation of subjects' work and activity impairment before and after treatment in both the investigational arm and the control arm. The Work Productivity and Activity Impairment (WPAI) questionnaire is a 6-question patient-reported general health assessment of productivity and activity impairment. WPAI results are expressed as the percentage of impairment from 0 to 100 where higher numbers indicate greater impairment or less productivity. Due to an error in the WPAI electronic data collection form, 2 questions were not visible to many subjects resulting in a significant amount of missing data for all scores except non-work activity impairment. Therefore, only the non-work activity impairment results are presented. As MM subjects were allowed to receive a crossover procedure after their 6-week follow-up visit, there is a limited number of MM subjects who completed the 12/24/52 visits.
Time Frame: 6,12,24,52 Week Follow-Up
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of Impairment
Arm/Group | Randomized ETBC | Randomized MM
Number analyzed (Participants) | 149 | 80
Percentage of Impairment
  Baseline: number analyzed (Participants) | 146 | 77
  Baseline | 45.3 (32.8) | 50.4 (31.1)
  6 Week Visit: number analyzed (Participants) | 141 | 70
  6 Week Visit | 16.6 (23.6) | 47.1 (32.0)
  12 Week Visit: number analyzed (Participants) | 133 | 11
  12 Week Visit | 10.9 (16.1) | 38.2 (27.5)
  24 Week Visit: number analyzed (Participants) | 130 | 8
  24 Week Visit | 12.0 (19.5) | 33.8 (37.0)
  52 Week Visit: number analyzed (Participants) | 124 | 4
  52 Week Visit | 9.1 (18.2) | 17.5 (20.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the procedure and at each follow-up visit at 2 weeks, 6 weeks, 12 weeks, 24 weeks, and 52 weeks post-treatment
Description: AEs in MM subjects prior to crossover are reported in the "Medical Management" arm (n=80). AEs in MM subjects after a crossover ETBC procedure are reported in the "Crossover MM" arm (n=70). To provide a robust safety profile, events are additionally presented in an "ALL ETBC" safety cohort, which consists of all subjects treated with the ETBC in the lead-in phase (n=80), randomized ETBC arm (n=149), and randomized MM arm who crossed over (n=70) for a total of 299 subjects in the "ALL ETBC" arm.
Groups:
- Lead-In: Subjects enrolled in the Lead-in group and treated with the ETBC
- Crossover MM: Subjects enrolled and randomized to treatment with Medical Management (MM) only who crossed over to have treatment with the ETBC after the 6-week follow-up visit
- ALL ETBC: All subjects in the lead-in phase, subjects randomized to the investigational arm who received treatment with the ETBC, and subjects in the control arm who crossed over to have treatment with the ETBC
- Randomized MM: Subjects enrolled and randomized to treatment with Medical Management (MM) only
Arm/Group | Lead-In | Randomized ETBC | Crossover MM | ALL ETBC | Randomized MM
All-Cause Mortality (participants affected / at risk) | 0/80 | 1/149 | 0/70 | 1/299 | 0/80
Serious Adverse Events (participants affected / at risk) | 2/80 | 5/149 | 0/70 | 7/299 | 1/80
Other Adverse Events (participants affected / at risk) | 30/80 | 58/149 | 20/70 | 108/299 | 18/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-In (N=80) | Randomized ETBC (N=149) | Crossover MM (N=70) | ALL ETBC (N=299) | Randomized MM (N=80)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-In (N=80) | Randomized ETBC (N=149) | Crossover MM (N=70) | ALL ETBC (N=299) | Randomized MM (N=80)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conductive deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 2 (3) | 2 (2) | 0 (0) | 4 (5) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 4 (4) | 1 (1) | 5 (5) | 1 (1)
Eustachian tube disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 3 (4) | 0 (0) | 3 (4) | 0 (0)
Eustachian tube obstruction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eustachian tube patulous (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 0 (0)
Otorrhea (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 4 (4) | 1 (1) | 5 (5) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Effusion (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myringitis bullous (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (4) | 4 (5) | 1 (1)
Otitis extrerna (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Otitis media (Infections and infestations) | 1 (2) | 4 (4) | 1 (1) | 6 (7) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 2 (4) | 7 (8) | 4 (4) | 13 (16) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 10 (11) | 6 (6) | 21 (23) | 0 (0)
Deafness traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days